CLINICAL TRIAL: NCT04992221
Title: Risk Factors Affected the Duration of Arterial Line Patency in ICU Bound COVID-19 Patients
Brief Title: Arterial Line Patency in ICU Bound COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-21-492
Record Dates: First submitted 2021-08-04; First posted 2021-08-05 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV-2 ICU Bound
Keywords: SARS-CoV-2; arterial line patency; Risk factors; ICU
MeSH Terms: interventions — Vascular Access Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: arterial line — arterial line inserted for invasice mointroing and sampling

SUMMARY:
The health care system was completely overwhelmed by the SARS-Cov-2 virus, and ICU admissions soared as a result of the ICU doctors' increased workload. A committed crew inserts invasive line procedures to guarantee a secure and efficient performance. When COVID-19 bound patients were followed up on in the second wave, frequent requests for arterial line placement were noted. These critically ill individuals had high rates of thrombosis, which was linked to thrombotic consequences. Many factors, such as patient morbidities, insertion technique, and operational health care trained personnel's qualifications, contribute to the lowering of arterial line patency.

Our ICU management committee approved the use of systemic anticoagulation of ICU admitted patients starting on March 21, 2021 in response to an increase in the incidence of thrombosis and pulmonary embolic events in patients with COVID-19 admitted to the ICU in the second wave of the epidemic.

DETAILED DESCRIPTION:
1. Introduction / Background The number of Coronavirus Disease 2019 (COVID-19) patients admitted to the intensive care unit has increased, and it has been noted that this pandemic is linked to high rates of thrombosis, which has exacerbated its effects on those critically ill patients.

In order to provide a multidisciplinary, safe service for invasive vascular procedures, as well as endotracheal intubations and the rapid response team (RRT) for quick assessment of deteriorating patients in the ward who were in need of ICU admission, which was reported before at a USA institute, we established a dedicated invasive procedure team from anesthetists during the peak admission of patients with COVID-19 to the ICU.

Invasive vascular access was employed for hemodynamic monitoring and management in patients undergoing high-risk surgery, especially in patients who were admitted to the intensive care unit.Different techniques, such as the use of heparinized fluids, are utilized to lower the incidence of arterial line failure.

Their main goal was to extend the average patency time of 5 to 10 days. When the arterial line was implanted for more than 2-3 days, the occlusion was documented. One frequent consequence is a transient arterial blockage.

We observed an upsurge in demand for arterial line insertions either in newly admitted or existing ICU patients during the COVID crisis. In addition to posing challenges for the ICU staff member, the repeated insertion of arterial lines raises the patient's risk for ischemia thrombosis and infectious occurrences in their limbs. However, there aren't many publications on the risk factors for arterial line blockages in ICU patients with COVID-19.

Our ICU management committee approved the use of systemic anticoagulation of ICU admitted patients starting on March 21, 2021 in response to an increase in the incidence of thrombosis and pulmonary embolic events in patients with COVID-19 admitted to the ICU in the second wave of this epidemic.

This observational study compares patients before and after the implementation of systemic anti coagulation to examine the effects of the medication on arterial line patency and the incidence of arterial line failure.

Identifying risk factors for impaired arterial line patency in both groups will be the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive ICU patients at HMGH Hospital; Hamad Medical Corporation with continuous invasive monitoring will be enrolled if they met following eligibility criteria: peripheral artery cannulation with a suitable arterial cannula and a functional arterial line established after insertion.

Exclusion Criteria:

* Other pateints with COVID-19 NOT ICU bound

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive ICU patients at HMGH Hospital; Hamad Medical Corporation with continuous invasive monitoring will be enrolled if they met following eligibility criteria: peripheral artery cannulation with a suitable arterial cannula and a functional arterial line established after insertion.
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of arterial line failure in ICU bound COVID-19 patients | 60-90 days

SECONDARY OUTCOMES:
Risk factors affecting the arterial line patency | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- HAMAD Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No